CLINICAL TRIAL: NCT04517214
Title: Phase II Study of Comparing Toripalimab Combined With GP Regimen Chemotherapy Versus GP Regimen Chemotherapy for Primary Metastatic Nasopharyngeal Carcinoma
Brief Title: Comparing Chemotherapy With/Without Toripalimab For Primary Metastatic Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Fudan University Eye and ENT Hospital (Unknown); Anhui Provincial Hospital (Other Government); Sir Run Run Shaw Hospital (Other); Hangzhou Cancer Hospital (Other); Ningbo Medical Center Lihuili Hospital (Other Government); The First People's Hospital of Changzhou (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Nanfang Hospital, Southern Medical University (Other); Shenzhen People's Hospital (Other); First Affiliated Hospital of Xi'anJiaotong Univerisity (Unknown); Guangzhou Panyu Central Hospital (Other); Fujian Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Chaosu Hu, Vice Director of Department of Radiation Oncology, Clinical Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRANSFORM
Record Dates: First submitted 2020-07-31; First posted 2020-08-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma; Primary metastatic; de novo metastatic; Toripalimab; PD-1; Immune checkpoint inhibitor; Chemotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab; Gemcitabine; Chemotherapy, Adjuvant; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Toripalimab Combined with GP Arm (Experimental): Systemic chemotherapy for 6 cycles: Toripalimab 240mg d1+Gemcitabine 1.0g/m2 d1, Cisplatin 80mg/m2 d1, q3w; Followed by Radiotherapy to the nasopharynx and neck; Then maintenance therapy of Toripalimab with Capecitabine: Toripalimab 240mg d1+Capecitabine 1000mg/m2 bid d1-14, q3w
  Interventions: Drug: Toripalimab; Radiation: IMRT to the nasopharynx and neck; Drug: Gemcitabine and Cisplatin Chemotherapy; Drug: Adjuvant chemotherapy with Capecitabine
- GP Arm (Active Comparator): Systemic chemotherapy for 6 cycles: Gemcitabine 1.0g/m2 d1, Cisplatin 80mg/m2 d1, q3w; Followed by Radiotherapy to the nasopharynx and neck; Then maintenance therapy of Capecitabine: Capecitabine 1000mg/m2 bid d1-14, q3w
  Interventions: Radiation: IMRT to the nasopharynx and neck; Drug: Gemcitabine and Cisplatin Chemotherapy; Drug: Adjuvant chemotherapy with Capecitabine

INTERVENTIONS:
Drug: Toripalimab — PD-1 inhibitor
  Other Names: JS001
  Arms: Toripalimab Combined with GP Arm
Radiation: IMRT to the nasopharynx and neck — IMRT to the nasopharynx and neck
  Other Names: RT to the nasopharynx and neck
Drug: Gemcitabine and Cisplatin Chemotherapy — Systemic chemotherapy
  Other Names: GP regimen chemotherapy
Drug: Adjuvant chemotherapy with Capecitabine — Adjuvant chemotherapy after radiation
  Other Names: Xeloda

SUMMARY:
The aim of this study is to compare the efficacy of Toripalimab Combined with GP Regimen Chemotherapy Versus GP Regimen Chemotherapy for Primary Metastatic NPC.

DETAILED DESCRIPTION:
About 4-10% of patients with nasopharyngeal carcinoma (NPC) have metastatic disease at diagnosis. The treatment recommendation of primary metastatic NPC is systemic chemotherapy. However, the optimal regimen is yet to determine due to lack of prospective randomized trial for this unique group of patients. Generally, GP regimen is used as the first-line treatment of primary metastatic NPC. The aim of this study is to compare the efficacy of Toripalimab Combined with GP Regimen Chemotherapy Versus GP Regimen Chemotherapy for Primary Metastatic NPC.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent;
2. Age older than 18 years old and younger than 70 years old;
3. Patients with newly histologically confirmed primary metastatic nasopharyngeal carcinoma;
4. At least one metastatic site that fulfills the criteria of "Evaluable Disease" per RECIST 1.1 Criteria;
5. Anticipated overall survival more than 3 months;
6. Satisfactory performance status: ECOG (Eastern Cooperative Oncology Group) scale 0-1;
7. No primary treatment of radiation, surgery, chemotherapy, targeted therapy and immune therapy post diagnosis of NPC;
8. Neutrophil ≥ 1.5×109 /L and PLT ≥100×109 /L and HGB ≥90 g/L;
9. With normal liver function test (ALT、AST ≤ 3×ULN, TBIL≤ 1.5×ULN, Albumin≥2.8g/dL );
10. With normal renal function test (Creatinine ≤ 1.5 ×ULN and creatinine clearance ≥60 ml/min);
11. HBV DNA<500 IU/mL（or 2500 copies/mL）and HCV RNA negative ;
12. Male and no pregnant female, able to adapt birth control methods during treatment.

Exclusion Criteria:

1. Hypersensitivity to Toripalimab, Gemcitabine, Cisplatin and Capecitabine;
2. Symptomatic spinal cord compression, or high-risk to develop pathological fracture that requires urgent surgery or radiation;
3. Necrotic disease, high-risk of massive nasal bleeding;
4. Suffered from malignant tumors, except cervical carcinoma in situ, papillary thyroid carcinoma, or skin cancer (non- melanoma) within five years;
5. Receive vaccine or live vaccine within 30 days prior to signing the informed consent;
6. Equivalent dose more than prednisone 10mg/d or other immunosuppressive treatments within 28 days prior to signing the informed consent;
7. Severe, uncontrolled medical conditions and infections;
8. Active, known or suspected autoimmune disease; Type I Diabetes, hypothyroidism those only need hormone replacement therapy; vitiligo or inactive asthma who don't need systemic therapy can recruit;
9. History of interstitial lung disease;
10. HIV positive;
11. Hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥500IU/ml, or 2500cps/ml; Positive HCV RNA;
12. Other diseases which may influence the safety or compliance of the clinical trial, such as heart failure with symptom, unstable angina, myocardial infarction, active infections those need systemic therapy, mental illness, or their family and society factors;
13. Women of child-bearing potential who are pregnant or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5 year
  PFS, defined as the time from randomization to the first documented objective tumor progression or death from any cause

SECONDARY OUTCOMES:
Objective Response Rate of Systemic chemotherapy | At the end of Cycle 6 of chemotherapy (each cycle is 21 days)
  ORR according to RECIST 1.1 Criteria
Disease Control Rate of Systemic chemotherapy | At the end of Cycle 6 of chemotherapy (each cycle is 21days)
  DCR according to RECIST 1.1 Criteria
The proportion of patients received radiotherapy to nasopharynx | 2 year
  Only patients with disease control after systemic chemotherapy will receive radiotherapy
Overall Survival | 5 year
  Defined from date of randomization to date of first documentation of death from Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
Progression-free Survival Rate | 1 year, 2 year rates
  Defined from date of randomization to date of first documentation of progression or death due to any cause.
Overall Survival Rate | 1 year, 2 year rates
  Defined from date of randomization to date of first documentation of death from Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
the Incidence of Adverse Effect | 1 year
  According to CTCAE 4.0.03
Changes of Quality of life, according to EORTC QLQ-C30 | 1 year
  According to EORTC QLQ-C30
Changes of Quality of life, according to EORTC QLQ-H&N35 | 1 year
  According to EORTC QLQ-H&N35

CONTACTS AND LOCATIONS:
Overall Officials: Chaosu Hu, M.D., Principal Investigator — Fudan University
Locations (1):
- Xiaomin Ou, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jiang F, Jin T, Feng XL, Jin QF, Chen XZ. Long-term outcomes and failure patterns of patients with nasopharyngeal carcinoma staged by magnetic resonance imaging in intensity-modulated radiotherapy era: The Zhejiang Cancer Hospital's experience. J Cancer Res Ther. 2015 Oct;11 Suppl 2:C179-84. doi: 10.4103/0973-1482.168181. PMID 26506872
- [Background] Ou X, Zhou X, Shi Q, Xing X, Yang Y, Xu T, Shen C, Wang X, He X, Kong L, Ying H, Hu C. Treatment outcomes and late toxicities of 869 patients with nasopharyngeal carcinoma treated with definitive intensity modulated radiation therapy: new insight into the value of total dose of cisplatin and radiation boost. Oncotarget. 2015 Nov 10;6(35):38381-97. doi: 10.18632/oncotarget.5420. PMID 26485757
- [Background] Lee AW, Ng WT, Chan LL, Hung WM, Chan CC, Sze HC, Chan OS, Chang AT, Yeung RM. Evolution of treatment for nasopharyngeal cancer--success and setback in the intensity-modulated radiotherapy era. Radiother Oncol. 2014 Mar;110(3):377-84. doi: 10.1016/j.radonc.2014.02.003. Epub 2014 Mar 11. PMID 24630534
- [Background] Lang J, Gao L, Guo Y, Zhao C, Zhang C; Society of Head & Neck Tumor Surgery; Society of Radiation Therapy; Chinese Anti-Cancer Association. Comprehensive treatment of squamous cell cancer of head and neck: Chinese expert consensus 2013. Future Oncol. 2014;10(9):1635-48. doi: 10.2217/fon.14.44. Epub 2014 Mar 17. PMID 24635574
- [Background] Chua MLK, Wee JTS, Hui EP, Chan ATC. Nasopharyngeal carcinoma. Lancet. 2016 Mar 5;387(10022):1012-1024. doi: 10.1016/S0140-6736(15)00055-0. Epub 2015 Aug 28. PMID 26321262
- [Background] Zou X, You R, Liu H, He YX, Xie GF, Xie ZH, Li JB, Jiang R, Liu LZ, Li L, Zhang MX, Liu YP, Hua YJ, Guo L, Qian CN, Mai HQ, Chen DP, Luo Y, Shen LF, Hong MH, Chen MY. Establishment and validation of M1 stage subdivisions for de novo metastatic nasopharyngeal carcinoma to better predict prognosis and guide treatment. Eur J Cancer. 2017 May;77:117-126. doi: 10.1016/j.ejca.2017.02.029. Epub 2017 Apr 7. PMID 28391025
- [Background] Sun XS, Liu LT, Liu SL, Guo SS, Wen YF, Xie HJ, Tang QN, Liang YJ, Li XY, Yan JJ, Ma J, Chen QY, Tang LQ, Mai HQ. Identifying optimal candidates for local treatment of the primary tumor among patients with de novo metastatic nasopharyngeal carcinoma: a retrospective cohort study based on Epstein-Barr virus DNA level and tumor response to palliative chemotherapy. BMC Cancer. 2019 Jan 21;19(1):92. doi: 10.1186/s12885-019-5281-5. PMID 30665378
- [Background] Chua DT, Sham JS, Au GK. A phase II study of docetaxel and cisplatin as first-line chemotherapy in patients with metastatic nasopharyngeal carcinoma. Oral Oncol. 2005 Jul;41(6):589-95. doi: 10.1016/j.oraloncology.2005.01.008. Epub 2005 Apr 14. PMID 15975521
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452